CLINICAL TRIAL: NCT03657498
Title: In Vivo Assessment of Natural Tooth Color, Pulp Vitality and Root Morphology After Combined Orthodontic-orthognathic Surgery Involving Maxillary Le Fort I Osteotomy
Brief Title: In Vivo Assessment of Natural Tooth Color After Orthognathic Surgery. A Pilot Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Konstantinos Lazaridis, Scientific assosiate, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 264/02.11.2010
Record Dates: First submitted 2018-07-16; First posted 2018-09-05 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Discoloration, Tooth
Keywords: Tooth color changes; Orthognathic surgery; Spectrophotometer
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Intervention Model Description: The trial includes a study group of patients receiving orthognathic surgery. It is divided into two subgroups. Subgroup I including bimaxillary surgical patients with Le-Fort I osteotomy for the upper jaw and sagittal split ramus osteotomy for the lower jaw. Subgroup II including patients receiving mandibular surgery only. Finally, two control groups were applied. Control group I including no treatment subjects and Control group II including standard orthodontic treatment subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group (Experimental): Combined orthodontic-orthognathic treatment
  Interventions: Procedure: Combined orthodontic-orthognathic treatment
- Control Group I (No Intervention): No intervention
- Control Group II (Active Comparator): Standard orthodontic treatment
  Interventions: Procedure: Standard orthodontic treatment

INTERVENTIONS:
Procedure: Combined orthodontic-orthognathic treatment — combined treatment including orthodontics and orthognathic surgery
  Arms: Study group
Procedure: Standard orthodontic treatment — treatment with standard orthodontic procedures
  Arms: Control Group II

SUMMARY:
In six consecutive patients planned to receive combined orthodontic-orthognathic surgery natural tooth color on 8 incisors was measured before initiation of the combined treatment (Time Point 1- baseline) and after its completion (Time Point 2- after intervention). The statistical interpretation of the results showed that tooth color change in the surgical group was higher in comparison to control groups. Control group I included non treatment subjects, while control group II included standard orthodontic treatment subjects. The results indicated that orthognathic surgery may affect natural tooth color but to small degree, as the color differences were just bellow the threshold value of 3.7 ΔΕ units. Under this value a color change cannot be easily detected by a human eye.

DETAILED DESCRIPTION:
The method of natural tooth color assessment included the use of the spectrophotometer Spectroshade Micro (MHT Zurich, Switzerland), which is a reflectance spectrophotometer with a LED technology light source with an output of 410-680 nm that is transformed into monochromatic light (λ = 400-720 nm) by means of grating. On this type of spectrophotometers, light is split so that teeth can be illuminated simultaneously from two sides at a 45° angle with the use of an intra-oral camera. The reflected light is directed at 0° on two detector areas (each detector area surface is of 18 x 13 mm2). One detector area is a color CCD chip responsible for the generation of the colored video image. A black-and-white CCD detector area records the spectrophotometric data. During a measuring process, light originating from the monochromator of the device is emitted in 10-nm intervals. Resulting images consist of 300,000 pixels. Initially, CIE tristimulus values are calculated and then converted to CIE-Lab values with the use of the accompanying software. Prior to every measuring cycle, the spectrophotometer had to be calibrated to a white and a green ceramic tile that are incorporated on the base of the device by the manufacturer.

Assessments were performed with closed lips in order to exclude disturbance by daylight. In order to avoid methodical errors in the assessment of luminance teeth of the upper and lower dental arches were not in contact, thereby obtaining a uniform black background by the oral cavity without an overlapping of anterior teeth. Tooth color was measured in the study and in the control groups at Time point 1 and Time Point 2. To enhance reliability of the method two sequential pictures of each tooth (Left + Right) were obtained with the use of the spectrophotometer and imported to the dedicated MHT Spectroshade software v3.01 Build 1007a (MHT Zurich, Switzerland), licensed to Aristotle University (Station ID: 952317337-Serial NR LUA164-164-164). Using the synchronization tool followed by the synchronous measurement tool, the cursor was accurately positioned on the center of the clinical crown on both pictures simultaneously, and the software reported color measurements for both pictures. The cursor shape was a circle, while the size was set at 100 pixels. Due to the synchronization of the pictures, the cursor area was exactly the same for both. To consider the method reliable, the maximal allowed color difference between the two consecutive pictures, was set at ΔΕ≤1.

ELIGIBILITY:
Inclusion Criteria:

* Absence of plaque accumulation and gingival inflammation. The Haemorrhagic index and Plaque index should be lower than 15 %.
* Absence of dental caries, prosthetic restorations, decalcifications, intrinsic and ⁄ or extrinsic discolorations, as well as morphologic ⁄ anatomical deviations in the measured teeth.
* Absence of severe crowding in the upper and lower dental arches (crowding should be lower than 4 mm).

Exclusion Criteria:

* Previous orthodontic treatment
* smoking
* previous bleaching procedure

Ages: 13 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2010-11-02 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Tooth color parameter L* change | Up to 49 months
  Lightness parameter of CIE-L*a*b* system
Tooth color parameter a* change | Up to 49 months
  Green-red component of CIE-L*a*b* system
Tooth color parameter b* change | Up to 49 months
  Blue-Yellow component of CIE-L*a*b* system

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Lazaridis, Dr, Principal Investigator — Aristotle University Of Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Karamouzos A, Athanasiou AE, Papadopoulos MA, Kolokithas G. Tooth-color assessment after orthodontic treatment: a prospective clinical trial. Am J Orthod Dentofacial Orthop. 2010 Nov;138(5):537.e1-8; discussion 537-9. doi: 10.1016/j.ajodo.2010.03.026. PMID 21055582